CLINICAL TRIAL: NCT03819153
Title: Effect of Semaglutide Versus Placebo on the Progression of Renal Impairment in Subjects With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: A Research Study to See How Semaglutide Works Compared to Placebo in People With Type 2 Diabetes and Chronic Kidney Disease
Acronym: FLOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4321; U1111-1217-6259 (Other: World Health Organization (WHO)); 2018-002878-50 (Registry Identifier: European Medicines Agency (EudraCT)); JapicCTI-194843 (Registry Identifier: JAPIC (Japan))
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants are to receive semglutide for up to 5 years or more (event driven). The trial is event driven with a pre-defined minimum number of renal endpoint events for the primary endpoint.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants are to receive placebo (semglutide) for up to 5 years or more (event driven). The trial is event driven with a pre-defined minimum number of renal endpoint events for the primary endpoint.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Participants are to inject semaglutide with a needle in the stomach, thigh or upper arm. Participants will use a pen to inject semaglutide under their skin. Participants will inject semaglutide 1 time a week on the same day of the week. Participants' dose of semaglutide will be changed over time. Participants start by taking a smaller amount (0.25 mg). After 4 weeks the dose will be increased to 0.5 mg. It will be increased more (to 1 mg) at 8 weeks. Participants will then stay on the same dose for the rest of the study.
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Participants are to inject placebo (semaglutide) with a needle in the stomach, thigh or upper arm. Participants will use a pen to inject placebo (semaglutide) under their skin. Participants will inject placebo (semaglutide) 1 time a week on the same day of the week. Participants' dose of placebo (semaglutide) will be changed over time. Participants start by taking a smaller amount (0.25 mg). After 4 weeks the dose will be increased to 0.5 mg. It will be increased more (to 1 mg) at 8 weeks. Participants will then stay on the same dose for the rest of the study.
  Arms: Placebo

SUMMARY:
The researchers are doing this study to see if semaglutide can slow down the growth and worsening of chronic kidney disease in people with type 2 diabetes. Participants will get semaglutide (active medicine) or placebo ('dummy medicine'). This is known as participants' study medicine - which treatment participants get is decided by chance. Semaglutide is a medicine, doctors can prescribe in some countries for the treatment of type 2 diabetes. Participants will get the study medicine in a pen. Participants will use the pen to inject the medicine in a skin fold once a week. The study will close when there is enough information collected to show clear result of the study. The total time participants will be in this study is about 3 to 5 years, but it could be longer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent. Japan: Male or female, age above or equal to 20 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus
* HbA1c less than or equal to 10% (less than or equal to 86 mmol/mol)
* Renal impairment defined either by:

  1. serum creatinine-based eGFR greater than or equal to 50 and less than or equal to 75 mL/min/1.73 m^2 (CKD-EPI) and UACR greater than 300 and less than 5000 mg/g or
  2. serum creatinine-based eGFR greater than or equal to 25 and less than 50 mL/min/1.73 m^2 (CKD-EPI) and UACR greater than 100 and less than 5000 mg/g
* Treatment with maximum labelled or tolerated dose of a renin-angiotensin-aldosterone system (RAAS) blocking agent including an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB), unless such treatment is contraindicated or not tolerated. Treatment dose must be stable for at least 4 weeks prior to the date of the laboratory assessments used for determination of the inclusion criteria for renal impairment and kept stable until screening

Exclusion Criteria:

* Congenital or hereditary kidney diseases including polycystic kidney disease, autoimmune kidney diseases including glomerulonephritis or congenital urinary tract malformations
* Use of any glucagon-like peptide-1 (GLP-1) receptor agonist within 30 days prior to screening
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 60 days prior to the day of screening
* Presently classified as being in New York Heart Association (NYHA) Class IV heart failure
* Planned coronary, carotid or peripheral artery revascularisation
* Current (or within 90 days) chronic or intermittent haemodialysis or peritoneal dialysis
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3533 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (411):
- United States (116):
  - Dr. Terence Hart, Tuscumbia, Alabama
  - California Inst Of Renal Res, Chula Vista, California
  - John Muir Physician Network, Concord, California
  - John Muir Physicians Network, Concord, California
  - Valley Research, Fresno, California
  - California Institute of Renal Research, La Mesa, California
  - First Valley Med Grp Lancaster, Lancaster, California
  - Clinical Trials Research_Sacramento, Lincoln, California
  - VA Loma Linda Hlthcr Sys, Loma Linda, California
  - Long Beach Center For Clinical Research, Long Beach, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Academic Medical Research Institute, Los Angeles, California
  - Valley Renal Medical Group Research, Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Saviers Medical Group, Port Hueneme, California
  - Inland Empire Clin Trials LLC, Rialto, California
  - Sierra Clinical Research, Roseville, California
  - California Research Foundation, San Diego, California
  - N America Res Inst - San Dimas, San Dimas, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - San Fernando Valley Hlth Inst, West Hills, California
  - Rocky Mount Reg VA Med-DN, Aurora, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - BayCare Medical Group - Endocrinology, Clearwater, Florida
  - Horizon Rs Grp, Coral Gbls, Coral Gables, Florida
  - Cesar Figueroa M.D. P.A., Delray Beach, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Palmetto Medical General Plaza, Hialeah, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - Homestead Associates In Research, Homestead, Florida
  - Life Spring Research, Miami, Florida
  - Oceane 7 Medical & Research Center, Inc., Miami, Florida
  - International Physicians Research, Miami, Florida
  - San Marcus Res Clin Miami Lakes, Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - South Broward Research LLC, Miramar, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - Cardiovascular Ctr of Sarasota, Sarasota, Florida
  - Clinical Research of Cent FL, Winter Haven, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Saltzer Medical Group Research, Nampa, Idaho
  - Apex Medical Research Inc, Chicago, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - North Suburban Nephrology LLC, Gurnee, Illinois
  - Endeavor Health, Skokie, Illinois
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - Metropolitan Cardiovascular Consultants, LLC, Beltsville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Elite Research Center, Flint, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University_St. Louis_0, St Louis, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Albany Medical College - Endo, Albany, New York
  - NYU Langone Neph Associates, Mineola, New York
  - NYU Nephrology Associates, New York, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - UNC Diabetes Care Center_Chapel Hill, Chapel Hill, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Eastern Nephr Assoc, PLLC, New Bern, North Carolina
  - Whiteville Medical Associates, Whiteville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Cincinnati Veterans Affairs Medical Center, Cincinnati, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Alliance for Multispec Res, Norman, Oklahoma
  - Heritage Valley Medical Group Inc, Beaver, Pennsylvania
  - Lycoming Internal Medicine, Inc., Jersey Shore, Pennsylvania
  - Northeast Endocrine Metabolic Associates, Philadelphia, Pennsylvania
  - Main Street Physician's Care, Little River, South Carolina
  - The Diabetes Center, LLC, Murrells Inlet, South Carolina
  - Family Medicine of SayeBrook LLC, Myrtle Beach, South Carolina
  - SC Nephrology and Hypertension, Orangeburg, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Vanderbilt Medical Center_Nashville, Nashville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Texas Diabetes & Endocrinology, P.A._Austin, Austin, Texas
  - Research Management, Inc, Austin, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Baylor Jack and Jane Hamilton, Dallas, Texas
  - Research Institute Of Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - MedResearch Inc, El Paso, Texas
  - Academy of Diabetes, T&E, El Paso, Texas
  - Juno Research, LLC_Houston, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Southwest Houston Research Ltd, Houston, Texas
  - Carlos Arauz-Pacheco Md, Pa, Rockwall, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Vermont Medical Center, South Burlington, Vermont
  - York Clinical Research LLC, Norfolk, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
  - MultiCare Inst for Res & Innov, Spokane, Washington
  - Universal Research Group, Tacoma, Washington
- Argentina (7):
  - Centro de Estudios Renales e Hipertensión Arterial, Villa Domínico, Buenos Aires
  - Centro Diabetológico y Nuticional Dr Alejandro Chertkoff, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - FEPREVA, CABA
  - Centro de Investigación Clínica, CABA
  - Glenny Corp. S.A, CABA
  - Medical Center of Diabetes and Nutrition, CABA
- Australia (8):
  - Gosford Renal Research, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital_Northmead, Westmead, New South Wales
  - Core Research Centre, Milton, Queensland
  - Monash Health Nephrology, Clayton, Victoria
  - St Vincent's Hospital_Fitzroy_0, Fitzroy, Victoria
  - Monash University Clinical Trial Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Belgium (9):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - Universitair Ziekenhuis Brussel - Diabeteskliniek, Brussels
  - UZ Brussel - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Gent - Endocrinologie - Diabetologie, Ghent
  - UZ Leuven - Endocrinology, Leuven
  - Centre hospitalier universitaire de Liège (CHU de Liège), Liège
  - AZ Delta - Roeselare, Roeselare
- Brazil (8):
  - Instituto de Ensino e Pesquisa Clínica do Ceará Ltda, Fortaleza, Ceará
  - Instituto Pró-Renal Brasil, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Dr. Christovão da Gama S.A., Santo André, São Paulo
  - Instituto de Pesquisa Clinica (IPEC), São Paulo, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Centro Médico Hospital da Bahia, Bahia
- Bulgaria (7):
  - Medical centre "Zdrave 1" OOD, Kozloduy
  - UMHAT "Kaspela", Depart. Endocrinology and Metab. Diseases, Plovdiv
  - MHAT "Dr. Ivan Seliminski"-Sliven, Sliven
  - "Nader Yabrudi - ASMPVBE Individual practice", Smolyan
  - UMHAT Aleksandrovska, Sofia
  - Medical Center Synexus Sofia, Sofia
  - Medical Center "Nov Rehabilitatsionen center" EOOD, Stara Zagora
- Canada (32):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - BC Diabetes Canada, Vancouver, British Columbia
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - QE II Health - Pharmacy, Halifax, Nova Scotia
  - Dr. Harpreet Bajaj, Brampton, Ontario
  - Aggarwal and Assoc Ltd., Brampton, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - LMC Clin Res Inc. Thornhill, Concord, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - Hamilton Med Res Group, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Milestone Research, London, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - King Street Research, Oshawa, Ontario
  - Bluewater Clin Res Group, Inc., Sarnia, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - Winterberry Family Medicine, Stoney Creek, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Dr Anil K Gupta Med Prof Corp, Toronto, Ontario
  - Dr. Anil K Gupta Med Prof Corp, Toronto, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Clinique de Recherche Medpharmgene Inc., Montreal, Quebec
  - Applied Med Inf Res, Montreal, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec
- China (5):
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital-Endocrinology, Beijing, Beijing Municipality
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'nan, Shandong
- France (14):
  - Centre Hospitalier Ardeche Nord, Annonay
  - Hospices Civils de Lyon-Hopital Cardiologique Louis Pradel-2, Bron
  - Centre Hospitalier Universitaire de Caen Normandie- Cote de Nacre-1, Caen
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-2, Grenoble - Cédex 09
  - Centre Hospitalier Departemental Vendee- La Roche Sur Yon, La Roche-sur-Yon
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-1, Le Creusot
  - Groupe SOS Santé Hôtel Dieu, Le Creusot
  - Fondation Rothschild, Paris
  - Centre Hospitalier Universitaire Reims-Hopital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Hôpital Nord Laënnec- Service D'Endocrinologie, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (9):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf
  - Medizinische Klinik 4, Universitätsklinikum Erlangen, Erlangen
  - InnoDiab Forschung GmbH, Essen
  - Praxis Dr. med. M. Esser, Essen
  - Wendisch/Dahl Hamburg, Hamburg
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
- Greece (13):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - Iatriko Psychicou Private Clinic, Athens
  - General hospital of Athens 'G.Gennimatas', Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - General Hospital of Athens "Laiko", Nephrology Clinic, Athens
  - General Hospital of Lamia, Lamia
  - General University Hospital of Patras,Nephrology clinic, Rio, Patra
  - AHEPA General University Hospital, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - Genl Hosp of Thessaloniki, Papageorgiou ,Nephrology clinic, Thessaloniki
- Hungary (13):
  - PTE-AOK II. Belgyogyaszati Klinika es Nephrologiai Centrum, Pécs, Baranya Vármegye
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Siófoki Kórház, Diabetológiai Szakrendelés, Siófok, Somogy County
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - Péterfy Sándor utcai Kórház, Budapest
  - MED-TIMA Kft., Budapest
  - Belinus Bt., Debrecen
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika D épület, Debrecen
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika, Debrecen
  - Békés Megyei Központi Kórház, Gyula
  - Siófoki Kórház, Diabetológiai Szakrendelés, Siófok
  - Markusovszky Egyetemi Oktatókórház, Szombathely
- India (17):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - BGS Global Hospitals, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Calicut Medical College, Kozhikode, Kerala
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Poona hospital and research centre, Pune, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Ajanta ResearchCentre, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Science, Lucknow, Uttar Pradesh
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Sir Ganga Ram Hospital, New Delhi
- Israel (4):
  - Diabetes Clinic Wolfson MC, Holon
  - Diabetes Unit Hadassah Ein Karem MC, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Kaplan Medical Center_Rehovot, Rehovot
- Italy (9):
  - Istituto Scientifico San Raffaele, Milan, MI
  - AOUPol.Giaccone UOC Malattie Endocrine,Ricambio e Nutrizione, Palermo, PA
  - Presidio Ospedaliero Cisanello, Pisa, PI
  - AO Papa Giovanni XXIII UOC malattie Endocrine 1-Diabetologia, Bergamo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale Maggiore Policlinico UO Endocrinologia Diabetolgia, Milan
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Roma
  - Azienda Ospedaliero - Universitaria Sant'Andrea, Roma
- Japan (27):
  - Seino Internal Medicine Clinic, Koriyama-shi, Fukushima, Japan
  - Manda Memorial Hospital, Sapporo-shi, Hokkaido, Hokkaido, Japan
  - Jinnouchi Hospital, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital, Miyazaki, Miyazaki
  - New Tokyo Heart Clinic, Chiba
  - Fukui Prefectural Hospital_Fukui, Fukui
  - Fukuoka Tokushukai Hospital, Fukuoka
  - Kawada Clinic, Gunma
  - Sasaki Hospital Internal Medicine, Hokkaido
  - Sasaki Internal Medicine, Hokkaido
  - Naka Kinen Clinic, Ibaraki
  - Nishiyamado Keiwa Hospital, Ibaraki
  - Kanazawa Medical University Hospital, Ishikawa
  - Yokohama Minoru Clinic, Kanagawa
  - H.E.C Science Clinic, Kanagawa
  - Shonan Takai Clinic, Kanagawa
  - Uji Tokushukai Medical Center, Kyoto
  - Kawasaki Medical School Hospital, Okayama
  - Takatsuki Red Cross Hospital, Osaka
  - Shimizu Clinic Fusa, Saitama
  - Oyama East Clinic, Tochigi
  - Tokyo Center Clinic, Tokyo
  - Fukuwa Clinic, Tokyo
  - Juntendo University Hospital_Tokyo, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Kato Clinic of Internal Medicine, Tokyo
  - Sugawara Clinic, Tokyo
- Malaysia (6):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak
  - Sarawak General Hospital, Kuching
  - Hospital Pulau Pinang, Pulau Pinang
  - Hospital Serdang, Serdang
- Mexico (6):
  - Centro de Atención al Diabetico, Actopan, Hidalgo
  - Inst. Jaliscience de Investigacion en Diabetes y Obesidad SC, Guadalajara, Jalisco
  - Instituto Nacional de Nutricion - Unidad de Inv de Enf Metab, Distrito Federal, México, D.F.
  - Instituto Nacional de Ciencias Médicas y Nutrición_Mexico City, Mexico City, México, D.F.
  - Centro para el Desarrollo de la Medicina y la Asistencia, Culiacán, Sinaloa
  - Centro de Estudios de Investigación Metabólicos y Cardio, Ciudad Madero, Tamaulipas
- Netherlands (9):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuis Groep Twente Almelo, Almelo
  - EB Flevo Research BV, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - OLVG West, Amsterdam
  - Amsterdam UMC Lokatie VUMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Tergooi, locatie Hilversum, Hilversum
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (8):
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik, Bialystok
  - NZOZ WITAMED Poradnia Diabetologiczna, Kielce
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Medyczne "Diabetika", Radom
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM W Szczecinie, Szczecin
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Miedzyleski Szpital Specjalistyczny, Oddzial Nefrologiczny, Warsaw
  - Prywatny Gabinet Janusz Gumprecht, Zabrze
- Russia (21):
  - Reg. State Budget Healthc. Inst. Regional Clinical Hospital, Barnaul
  - City Hospital #5, Barnaul
  - Road Clinical Hospital at station Chelyabinsk, Chelyabinsk
  - PIH "Clin Hosp "RZD-Medicina" former Kazan OJSC Rus Railways, Kazan'
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - National Medical Research Center of Endocrinology, Moscow
  - LLC RC Medical, Novosibirsk
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Joint Stock Company "Modern Medical Technologies", Saint Petersburg
  - Aurora MedFort LLC, Saint Petersburg
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - Medinet LLC, Saint Petersburg
  - LLC "Endocrinolog", Samara
  - SHI Saratov City Clinical Hospital #9, Saratov
  - Regional clinical cardiology dispensary, Saratov
  - Regional Endocrinological Dispensary, Stavropol
  - Ulianovsk Regional Clinical Hospital, Ulyanovsk
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - Solovyev Clinical Emergency Hospital, Yaroslavl
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Slovakia (10):
  - MEDISPEKTRUM s.r.o., Bratislava
  - FMC - dialyzacne sluzby, s.r.o., Košice
  - IN-DIA s.r.o., Lučenec
  - Narodny Endokrinologicky a diabetologicky ustav, Ľubochňa
  - DIABETIK s.r.o., Nitra
  - Diabetologicka ambulancia MEDIKARD, s.r.o., Prešov
  - ARETEUS s.r.o., Trebišov
  - MUDr. Jana Rociakova s.r.o., ambulancia vnutorneho lekarstva, Žilina
  - FMC- dialyzacne sluzby, s.r.o., Žilina
  - MEDIVASA, s.r.o., Diabetologicka ambulancia, Žilina
- South Africa (9):
  - Diabetes Care Centre & CDE Centre, Benoni, Gauteng
  - LCS Clinical Research Unit, Cosmo City, Gauteng
  - Soweto Clinical Trial Centre, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Dr A Amod, Durban, KwaZulu-Natal
  - Precise Clinical Solutions (Pty) Ltd, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Prof Rayner_Division of Nephrology, Cape Town, Western Cape
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Público da Mariña, Burela de Cabo
  - Hospital Universitario de Getafe, Getafe
  - Hospital Ribera Polusa, Lugo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
- Thailand (7):
  - Siriraj Hospital_Bangkoknoi, Bangkok, Bangkoknoi, Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Mueang Chiang Mai District
  - Phramongkutklao Hospital-nephrology, Bangkok, Rajathewee
  - King Chulalongkorn Memorial Hospital-Division of Nephrology, Bangkok
  - King Chulalongkorn Memorial Hospital_Bangkok, Bangkok
  - Phramongkutklao Hospital-nephrology, Bangkok
  - Siriraj Hospital-Nephro, Bangkok
- Turkey (Türkiye) (12):
  - Ankara Universitesi Ibni Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Nefroloji Bilim Dali, Ankara
  - Gazi University Medical Faculty- Nephrology, Ankara
  - Akdeniz Universitesi Hastanesi Nefroloji Bilim Dali, Antalya
  - Aydin Adnan Menderes University Nephrology, Aydin
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi- Nefroloji, Istanbul
  - Goztepe Egitim Arastirma Hastanesi Nefroloji, Istanbul
  - T.C. Saglik Bakanligi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş
  - Kocaeli University Nephrology Department, Kocaeli
- Ukraine (7):
  - SI "Institute of Medical and Social Problems of Disability", Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - CNPI "Kharkiv City Clinical Hospital #27", Kharkiv
  - SI "National Institute of Therapy n.a. L.T. Malaya of NAMSU", Kharkiv
  - Institute of Endocrinology and Metabolism of AMSU, Kyiv
  - CI "1st City Clinical Hospital of Poltava City Council", Poltava
  - CI "Zaporizhia city clinical hospital #10", Zaporizhia
- United Kingdom (11):
  - Aberdeen Royal Infirmary, Aberdeen
  - Diabetes Centre, Heartlands Hospital, Birmingham, Birmingham
  - Ely Bridge Surgery, Cardiff
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Glasgow Clinical Research Facility, Glasgow
  - The Diabetes Centre, Ipswich
  - North Middlesex Hospital, London
  - Royal Free - Diabetes, London
  - Lister Hospital, Stevenage
  - St Georges Hospital, Tooting

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Background] Rossing P, Baeres FMM, Bakris G, Bosch-Traberg H, Gislum M, Gough SCL, Idorn T, Lawson J, Mahaffey KW, Mann JFE, Mersebach H, Perkovic V, Tuttle K, Pratley R. The rationale, design and baseline data of FLOW, a kidney outcomes trial with once-weekly semaglutide in people with type 2 diabetes and chronic kidney disease. Nephrol Dial Transplant. 2023 Aug 31;38(9):2041-2051. doi: 10.1093/ndt/gfad009. PMID 36651820
- [Derived] Rossing P, Lindhardt M, Tikkanen CK, Menon J, Cattin J, Hunt B, Malkin SJP, Chubb B, Damgaard T, Borg R. Once-weekly semaglutide versus placebo for the treatment of type 2 diabetes and chronic kidney disease in Denmark: A long-term cost-effectiveness analysis based on FLOW. Cardiovasc Diabetol. 2025 Dec 20. doi: 10.1186/s12933-025-03002-1. Online ahead of print. PMID 41422027
- [Derived] Pruijm M, Belmar N, Bjornstad P, Cherney DZI, Das V, Gunnarsson T, Hodgin JB, Schytz PA, Tuttle KR, Kretzler M. REMODELing mechanistic trials for kidney disease: a multimodal, tissue-centered approach to understand the renal mechanism of action of semaglutide. Kidney Int. 2026 Jan;109(1):6-16. doi: 10.1016/j.kint.2025.10.005. Epub 2025 Nov 7. PMID 41207620
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Mendonca L, Moura H, Chaves PC, Neves JS, Ferreira JP. The Impact of Glucagon-Like Peptide-1 Receptor Agonists on Kidney Outcomes: A Meta-Analysis of Randomized Placebo-Controlled Trials. Clin J Am Soc Nephrol. 2024 Oct 8;20(2):159-68. doi: 10.2215/CJN.0000000584. Online ahead of print. PMID 39480988
- [Derived] Kosiborod MN, Deanfield J, Pratley R, Borlaug BA, Butler J, Davies MJ, Emerson SS, Kahn SE, Kitzman DW, Lingvay I, Mahaffey KW, Petrie MC, Plutzky J, Rasmussen S, Ronnback C, Shah SJ, Verma S, Weeke PE, Lincoff AM; SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM Trial Committees and Investigators. Semaglutide versus placebo in patients with heart failure and mildly reduced or preserved ejection fraction: a pooled analysis of the SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM randomised trials. Lancet. 2024 Sep 7;404(10456):949-961. doi: 10.1016/S0140-6736(24)01643-X. Epub 2024 Aug 30. PMID 39222642
- [Derived] Pratley RE, Tuttle KR, Rossing P, Rasmussen S, Perkovic V, Nielsen OW, Mann JFE, MacIsaac RJ, Kosiborod MN, Kamenov Z, Idorn T, Hansen MB, Hadjadj S, Bakris G, Baeres FMM, Mahaffey KW; FLOW Trial Committees and Investigators. Effects of Semaglutide on Heart Failure Outcomes in Diabetes and Chronic Kidney Disease in the FLOW Trial. J Am Coll Cardiol. 2024 Oct 22;84(17):1615-1628. doi: 10.1016/j.jacc.2024.08.004. Epub 2024 Aug 30. PMID 39217553
- [Derived] Mann JFE, Rossing P, Bakris G, Belmar N, Bosch-Traberg H, Busch R, Charytan DM, Hadjadj S, Gillard P, Gorriz JL, Idorn T, Ji L, Mahaffey KW, Perkovic V, Rasmussen S, Schmieder RE, Pratley RE, Tuttle KR. Effects of semaglutide with and without concomitant SGLT2 inhibitor use in participants with type 2 diabetes and chronic kidney disease in the FLOW trial. Nat Med. 2024 Oct;30(10):2849-2856. doi: 10.1038/s41591-024-03133-0. Epub 2024 Jun 24. PMID 38914124
- [Derived] De La Flor JC, Moral E, Deira J, Monzon T, Valga F, Albarracin C, Rodeles M. Response to "Experience with dulaglutide in an obese diabetic patient on incremental peritoneal dialysis". Response to related letter. Nefrologia (Engl Ed). 2024 May-Jun;44(3):444-446. doi: 10.1016/j.nefroe.2023.10.010. Epub 2024 Jun 10. No abstract available. PMID 38862303
- [Derived] Perkovic V, Tuttle KR, Rossing P, Mahaffey KW, Mann JFE, Bakris G, Baeres FMM, Idorn T, Bosch-Traberg H, Lausvig NL, Pratley R; FLOW Trial Committees and Investigators. Effects of Semaglutide on Chronic Kidney Disease in Patients with Type 2 Diabetes. N Engl J Med. 2024 Jul 11;391(2):109-121. doi: 10.1056/NEJMoa2403347. Epub 2024 May 24. PMID 38785209
- [Derived] Cohen S, Sternlicht H, Bakris GL. Mineralocorticoid Receptor Antagonists in the Treatment of Diabetic Kidney Disease: Their Application in the Era of SGLT2 Inhibitors and GLP-1 Receptor Agonists. Curr Diab Rep. 2022 May;22(5):213-218. doi: 10.1007/s11892-022-01461-4. Epub 2022 Apr 20. PMID 35441935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were randomized to treatment at 383 sites in 28 countries as follows: Argentina (7); Australia (7); Belgium (8); Brazil (7); Bulgaria (7); Canada (25); China (4); France (11); Germany (9); Greece (13); Hungary (10); India (16); Israel (4); Italy (8); Japan (26); Malaysia (6); Mexico (6); Netherlands (9); Poland (7); Russia (21); Slovakia (10); South Africa (8); Spain (7); Thailand (6); Turkey (12); Ukraine (7); United Kingdom (11); and United States (111).
Pre-assignment Details: A total of 3533 eligible participants were randomized (1:1) to treatment with semaglutide 1 milligram (mg) (1767) or placebo (1766). The study included a treatment period (up to 60 months or more) and a follow-up period (5 weeks).
Groups:
- Semaglutide: Participants received a dose of semaglutide subcutaneously once weekly with dose escalation in every 4 weeks in doses 0.25 mg (weeks 0-3), 0.50 mg (weeks 4-7) until the maintenance dose of 1 mg was reached at week 8 and continued 1 mg dose along with standard of care until end of the study (week 238). Participants were followed up for 5 weeks after end of treatment.
- Placebo: Participants received placebo matching semaglutide subcutaneously once weekly along with standard of care until end of the study (week 238). Participants were followed up for 5 weeks after end of treatment.
Period: Overall Study
Arm/Group | Semaglutide | Placebo
Started | 1767 | 1766
Full Analysis Set (FAS) | 1767 | 1766
Completed | 1724 | 1708
Not Completed | 43 | 58
Not completed — Withdrawal by Subject | 20 | 28
Not completed — Lost to Follow-up | 23 | 30

BASELINE CHARACTERISTICS:
Population: Analysis of participants were performed on full analysis set (FAS) that was defined as all unique randomised participants and were grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Placebo | Total
Number analyzed (Participants) | 1767 | 1766 | 3533
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (9.0) | 66.7 (9.0) | 66.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519 | 550 | 1069
  Male | 1248 | 1216 | 2464
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 273 | 283 | 556
  Not Hispanic or Latino | 1421 | 1411 | 2832
  Unknown or Not Reported | 73 | 72 | 145
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 9 | 16 | 25
  Race: Asian | 439 | 407 | 846
  Race: Black or African American | 78 | 82 | 160
  Race: Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Race: White | 1155 | 1168 | 2323
  Race: Other | 45 | 50 | 95
  Race: Not reported | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Time of Randomization to First Occurrence of Onset of Persistent ≥50% Reduction in eGFR(CKD-EPI); Onset of Persistent eGFR(CKD-EPI) <15mL/Min/1.73m^2; Initiation of Chronic Renal Replacement Therapy; Renal Death; CV Death
Description: Number of participants with first composite renal event i.e., from time of randomization to first occurrence of an onset of persistent greater than or equal to (≥) 50 percent (%) reduction in estimated glomerular filtration rate (eGFR) (chronic kidney disease - epidemiology collaboration [CKD-EPI]), onset of persistent eGFR (CKD-EPI) <15 milliliter per minute per 1.73 meter square (mL/min/1.73m^2), initiation of chronic renal replacement therapy (dialysis or kidney transplantation), renal death, and cardiovascular (CV) death combined data were reported in this outcome measure.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 331 | 410
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Time from randomization to first composite renal event was analyzed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by use of sodium glucose cotransporter-2 (SGLT-2) inhibitor (yes/no) at baseline. Based on the available number of events for analysis, the nominal significance level was updated to 0.01612 using the Lan-DeMets alpha spending function. eGFR was calculated using the CKD-EPI formula; Test type: Superiority; p = 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.66 to 0.88]

2. Secondary Outcome: Annual Rate of Change in eGFR (CKD-EPI) (Total eGFR Slope)
Description: Annual rate of change in Total eGFR slope CKD-EPI were reported from baseline at Week 234 in-trial period. eGFR was calculated using the CKD-EPI formula. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: (mL/min/1.73 m^2)/year
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
(mL/min/1.73 m^2)/year | -2.19 (0.1) | -3.36 (0.1)

3. Secondary Outcome: Number of Participants From Time of Randomization to Occurrence of Onset of Persistent ≥50% Reduction in eGFR (CKD-EPI)
Description: Number of participants from time of randomization to time to occurrence of onset of persistent ≥50% reduction in eGFR (CKD-EPI) were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 165 | 213

4. Secondary Outcome: Number of Participants From Time of Randomization to Occurrence of Onset of Persistent eGFR (CKD-EPI) <15mL/Min/1.73m^2
Description: Number of participants from time of randomization to time to occurrence of onset of persistent eGFR (CKD-EPI) <15 mL/min/1.73m^2 were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 92 | 110

5. Secondary Outcome: Number of Participants From Time of Randomization to Occurrence of Initiation of Chronic Renal Replacement Therapy
Description: Number of participants from time of randomization to time to occurrence of initiation of chronic renal replacement therapy (dialysis or kidney transplantation) were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 87 | 100

6. Secondary Outcome: Number of Participants From Time of Randomization to Occurrence of Renal Death
Description: Number of participants from time of randomization to time to occurrence of renal death were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 5 | 5

7. Secondary Outcome: Number of Participants From Time of Randomization to Occurrence of CV Death
Description: Number of participants from time of randomization to time to occurrence of CV death were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 123 | 169

8. Secondary Outcome: Annual Rate of Change in eGFR (Chronic Kidney Disease CKD-EPI) (Chronic eGFR Slope)
Description: Annual rate of change in eGFR in terms of chronic kidney disease CKD-EPI were reported from Week 12 to Week 234 in-trial period. eGFR was calculated using the CKD-EPI formula. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Week 12, Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization. Here 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1735 | 1736
mL/min/1.73 m^2 | -2.36 (0.1) | -3.30 (0.1)

9. Secondary Outcome: Change From Baseline in eGFR (CKD-EPI) at Week 12
Description: Change from baseline in eGFR at Week 12 during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1665 | 1663
mL/min/1.73m^2 | -1.07 (8.16) | -1.07 (7.73)

10. Secondary Outcome: Change From Baseline in eGFR (Cystatin C CKD-EPI) at Week 104
Description: Changes from baseline in eGFR (cystatin C) at Week 104 in-trial period were reported. Cystatin C was calculated using the CKD-EPI formula. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1425 | 1391
mL/min/1.73m^2 | -2.1 (11.4) | -5.4 (9.7)

11. Secondary Outcome: Change From Baseline in Urinary Albumin-to-creatinine Ratio (UACR) at Week 104: Ratio to Baseline
Description: Change from baseline in UACR (ratio to baseline) at Week 104 in-trial period were reported. For UACR, the baseline assessment is defined as the mean of the two assessments from the randomization visit. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1454 | 1423
Ratio | 0.60 (224.09) | 0.89 (211.70)

12. Secondary Outcome: Number of Participants From Time of Randomization to Time to First Occurrence of a Major Adverse Cardiovascular Event (MACE): Acute Myocardial Infarction (Non Fatal); Non-fatal Stroke; and CV Death
Description: Number of participants who reported first occurence of non-fatal acute myocardial infarction, non-fatal stroke, and CV death combined data were presented from Week 0 up to Week 234 during on-treatment period. MACE consisted of non-fatal acute myocardial infarction, cardiovascular death and non-fatal stroke. First on-treatment period is defined as period from date of first dose until first time where no dose had been administered within 5 weeks (35 days) or end of the in-trial period, whichever came first.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 212 | 254

13. Secondary Outcome: Number of Participants From Time of Randomization to Time to Occurrence of All-cause Death
Description: Number of participants who reported occurence of deaths from Week 0 up to Week 234 during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 227 | 279

14. Secondary Outcome: Number of Participants From Time of Randomization to Time to Occurrence of Each of the Individual Components of the Confirmatory Secondary MACE Endpoint: Non-fatal Myocardial Infarction
Description: Number of participants who reported occurrence of non-fatal acute myocardial infarction from Week 0 up to Week 234 during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 52 | 64

15. Secondary Outcome: Number of Participants From Time of Randomization to Time to Occurrence of Each of the Individual Components of the Confirmatory Secondary MACE Endpoint: Non-fatal Stroke
Description: Number of participants who reported occurrence of non-fatal stroke from Week 0 up to Week 234 during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 63 | 51

16. Secondary Outcome: Number of Participants From Time of Randomization to Time to First Occurrence of Major Adverse Limb Events (MALE): Acute Limb Ischaemia Hospitalization and Chronic Limb Ischaemia Hospitalization
Description: Number of participants with combined data of first occurence of acute limb ischaemia hospitalization and chronic limb ischaemia hospitalization from Week 0 up to Week 234 during on-treatment period were presented. MALE consisted of acute and chronic limb ischaemia hospitalisation.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants | 16 | 28

17. Secondary Outcome: Number of Participants With Acute Limb Ischaemia Hospitalization and Chronic Limb Ischaemia Hospitalization
Description: Number of participants of acute limb ischaemia hospitalization and chronic limb ischaemia hospitalization from Week 0 up to Week 234 during in-trial period were presented. MALE consisted of acute and chronic limb ischaemia hospitalisation. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Participants
  Acute limb ischaemia hospitalization | 1 | 3
  Chronic limb ischaemia hospitalization | 16 | 25

18. Secondary Outcome: Change From Baseline in Body Weight at Week 104
Description: Change in body weight from Week 0 up to Week 104 during in-trial period, measured in kilograms, were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baeline (Week 0), Week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1502 | 1468
Kilograms | -5.54 (6.57) | -1.43 (6.33)

19. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) at Week 104
Description: Change in HbA1c from Week 0 to Week 104 during in-trial period, measured in percentage point of HbA1c, were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1448 | 1427
Percentage of HbA1c | -0.86 (1.35) | -0.04 (1.29)

20. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 104
Description: Change in systolic blood pressure from Week 0 to Week 104 during in-trial period were presented. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1511 | 1472
Millimeters of mercury | -3.9 (17.6) | -1.4 (18.3)

21. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 104
Description: Change in diastolic blood pressure from Week 0 to Week 104 during in-trial period were reported. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: Baseline (Week 0), Week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1511 | 1472
millimeters of mercury | -0.4 (9.6) | -0.8 (10.4)

22. Secondary Outcome: Number of Severe Hypoglycaemic Episodes
Description: The number of severe hypoglycaemic episodes (such as the seriousness of hypoglycaemia, contributing factors, seizures, and unconsciousness; classified by American Diabetes Association) observed during the in-trial period were reported in this endpoint. In-trial observation period was defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death.
Time Frame: From Week 0 up to Week 234
Population: FAS included all unique randomized participants who were grouped according to the treatment assigned at randomization.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1767 | 1766
Episodes | 37 | 37

ADVERSE EVENTS:
Time Frame: From Week 0 up to Week 238
Description: The safety evaluation was based on the FAS using the in-trial observation period which is defined as the period from date of randomization to the first of (both inclusive): date of follow-up visit, date when participant withdrew consent, date of last contact with participant (for participant lost to follow-up), and date of death. Details on the approach followed for collecting the AEs is mentioned in the section 9.3 of protocol.
Arm/Group | Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 227/1767 | 279/1766
Serious Adverse Events (participants affected / at risk) | 877/1767 | 950/1766
Other Adverse Events (participants affected / at risk) | 507/1767 | 522/1766
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=1767) | Placebo (N=1766)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 4 (4) | 2 (3)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 5 (5) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 124 (165) | 123 (143)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 6 (6)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 49 (52) | 67 (81)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (13)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 32 (37)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 18 (25) | 24 (28)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 13 (16) | 16 (16)
Angina unstable (Cardiac disorders) | 12 (12) | 22 (24)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 4 (4)
Aortic aneurysm rupture (Vascular disorders) | 4 (4) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (2)
Aortic stenosis (Vascular disorders) | 7 (7) | 2 (2)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 3 (3)
Aortoenteric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 8 (8) | 5 (5)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 3 (3) | 3 (3)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 2 (2)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 4 (7) | 5 (5)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 31 (35) | 22 (31)
Atrial flutter (Cardiac disorders) | 11 (14) | 7 (10)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (6) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 5 (5) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 4 (4) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 4 (4) | 3 (3)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Bacteraemia (Infections and infestations) | 3 (3) | 5 (5)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Behcet's syndrome (Vascular disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1) | 1 (1)
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 4 (4)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood folate decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 2 (2)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 2 (2)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 6 (7) | 6 (6)
Brain compression (Nervous system disorders) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 2 (2) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 58 (59) | 74 (74)
COVID-19 pneumonia (Infections and infestations) | 68 (68) | 83 (83)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 16 (18) | 14 (14)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 48 (63) | 66 (89)
Cardiac failure acute (Cardiac disorders) | 27 (30) | 26 (32)
Cardiac failure chronic (Cardiac disorders) | 18 (19) | 18 (19)
Cardiac failure congestive (Cardiac disorders) | 33 (40) | 49 (56)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pacemaker removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 6 (6)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 3 (3)
Cardiorenal syndrome (Cardiac disorders) | 3 (3) | 3 (3)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 2 (2) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 7 (8) | 3 (3)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 22 (27) | 13 (16)
Cataract operation (Surgical and medical procedures) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 12 (17) | 26 (31)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Central cord syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral cyst (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 4 (4)
Cerebral infarction (Nervous system disorders) | 11 (12) | 5 (5)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 15 (15) | 13 (13)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Chagas' cardiomyopathy (Infections and infestations) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 9 (9) | 5 (5)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholangitis infective (Infections and infestations) | 1 (2) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 12 (12) | 15 (16)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 13 (13) | 12 (12)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestatic liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chorioretinitis (Infections and infestations) | 0 (0) | 1 (1)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 42 (48) | 37 (37)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 9 (10)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 3 (3)
Claudication of jaw muscles (Vascular disorders) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 3 (4) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (6)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Contrast media toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (2)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 31 (37) | 28 (29)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 8 (11) | 10 (11)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 2 (2)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cranial nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Craniofacial fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (General disorders) | 21 (21) | 30 (30)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 10 (13) | 10 (10)
Delirium (Psychiatric disorders) | 4 (4) | 3 (3)
Dementia (Nervous system disorders) | 4 (4) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 1 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 4 (5)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Diabetic autonomic neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic complication renal (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic end stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 11 (14) | 12 (12)
Diabetic foot infection (Infections and infestations) | 6 (8) | 7 (8)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 10 (12) | 7 (9)
Diabetic macroangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Diabetic nephropathy (Renal and urinary disorders) | 9 (12) | 5 (6)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Diabetic retinal oedema (Eye disorders) | 3 (4) | 1 (1)
Diabetic retinopathy (Eye disorders) | 12 (15) | 9 (9)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 4 (4)
Dilatation intrahepatic duct congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 11 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 1 (1)
Encephalomalacia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 7 (8) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 31 (33) | 36 (37)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 7 (8) | 3 (3)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Exfoliation glaucoma (Eye disorders) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 17 (18) | 20 (21)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Flatback syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (2)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 10 (14) | 11 (12)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (8) | 6 (6)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (9) | 10 (10)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
General symptom (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 4 (4)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glomerular filtration rate abnormal (Investigations) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 2 (2)
Glomerulonephritis proliferative (Renal and urinary disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 4 (4)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 4 (4) | 5 (5)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 3 (4)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (3) | 4 (4)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (11) | 11 (15)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (18) | 23 (24)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperplasia (General disorders) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 9 (13) | 17 (19)
Hypertensive crisis (Vascular disorders) | 7 (10) | 7 (7)
Hypertensive emergency (Vascular disorders) | 4 (4) | 4 (4)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 8 (8) | 6 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 4 (4) | 15 (19)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 22 (23) | 24 (27)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 14 (16) | 7 (7)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 4 (5)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infective aortitis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 3 (3)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 2 (2)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (6)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 23 (23) | 34 (36)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lacunar infarction (Nervous system disorders) | 0 (0) | 3 (3)
Lacunar stroke (Nervous system disorders) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 8 (10)
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular failure (Cardiac disorders) | 5 (6) | 11 (11)
Leg amputation (Surgical and medical procedures) | 2 (2) | 0 (0)
Leriche syndrome (Vascular disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Linear IgA disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 2 (3)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 3 (3)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 2 (2)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 3 (3) | 0 (0)
Macular oedema (Eye disorders) | 2 (3) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (4)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (3) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Metabolic encephalopathy (Nervous system disorders) | 5 (5) | 3 (4)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 5 (5) | 2 (2)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucosal hypertrophy (General disorders) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 9 (9)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelodysplastic syndrome with single lineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 15 (15) | 15 (15)
Myocardial ischaemia (Cardiac disorders) | 10 (10) | 3 (3)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 2 (2)
Necrotising oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 7 (7) | 5 (5)
Nephropathy (Renal and urinary disorders) | 2 (2) | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (2)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 8 (8)
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ocular ischaemic syndrome (Eye disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 4 (4)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (3) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 3 (3)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
Osteomyelitis (Infections and infestations) | 9 (11) | 13 (15)
Osteomyelitis acute (Infections and infestations) | 3 (3) | 1 (1)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pacing induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 5 (5)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Parapharyngeal space infection (Infections and infestations) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Penile abscess (Infections and infestations) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pericardial calcification (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2) | 4 (4)
Pericarditis uraemic (Cardiac disorders) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 10 (11) | 19 (29)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 3 (3) | 4 (4)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 9 (9)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 3 (3)
Peripheral vascular haematoma (Vascular disorders) | 0 (0) | 1 (1)
Peritoneocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 7 (7)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (6)
Pleurisy viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 66 (70) | 75 (87)
Pneumonia aspiration (Infections and infestations) | 6 (7) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 3 (4) | 11 (11)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 5 (5) | 3 (3)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Primary amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 6 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Prosthetic cardiac valve malfunction (Product Issues) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Pseudoaneurysm infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudohypoaldosteronism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 14 (14)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Pulse abnormal (Investigations) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 5 (5) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 4 (6)
Pyelonephritis chronic (Infections and infestations) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 7 (7)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 4 (5)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 8 (8) | 17 (17)
Renal impairment (Renal and urinary disorders) | 9 (9) | 18 (21)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal transplant (Surgical and medical procedures) | 0 (0) | 2 (2)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 11 (12)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (2) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
SARS-CoV-2 sepsis (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 3 (3) | 3 (3)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 17 (20) | 23 (24)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Septic pulmonary embolism (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 8 (8) | 14 (14)
Serous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 2 (2)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Skin lesion removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (13)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (6) | 2 (2)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 3 (3)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 3 (3)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 2 (2)
Subcapsular renal haematoma (Renal and urinary disorders) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 5 (7)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 4 (4) | 3 (3)
Sudden death (General disorders) | 5 (5) | 10 (10)
Suicide attempt (Psychiatric disorders) | 0 (0) | 3 (4)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 14 (16) | 9 (9)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 1 (1)
Thalamic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tidal volume decreased (Investigations) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 3 (3)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tractional retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 15 (15) | 13 (14)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (6)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 2 (2) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 2 (3)
Upper motor neurone lesion (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Uraemic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 3 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (7) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 23 (27) | 27 (30)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 3 (3) | 3 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 3 (3)
Vascular device infection (Infections and infestations) | 2 (2) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular shunt (Vascular disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vasculitis necrotising (Vascular disorders) | 1 (1) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (11) | 5 (5)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=1767) | Placebo (N=1766)
COVID-19 (Infections and infestations) | 221 (238) | 246 (260)
Diabetic retinopathy (Eye disorders) | 339 (394) | 325 (381)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03819153/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT03819153/SAP_001.pdf